CLINICAL TRIAL: NCT04870996
Title: A Randomised Controlled Trial of Concurrent Cognitive Training and Transcranial Direct Current Stimulation or Cognitive Training Alone in Patients With Schizophrenia.
Brief Title: RCT of tDCS Combined With Cognitive Training in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHAN SAU MAN, SANDRA (Other)
Responsible Party: Sponsor-Investigator, CHAN SAU MAN, SANDRA, Associate Professor, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CRE-2019.239
Record Dates: First submitted 2021-04-22; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Schizophrenia
Keywords: cognitive training; transcranial direct current stimulation; cognitive intervention; cognitive dysfunction; schizophrenia
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active transcranial Direct Current Stimulation (tDCS) + Cognitive training (CT) (Experimental): Twenty-three participants received five treatment sessions of concurrent active tDCS and CT on five consecutive days. The participants received a ramp-up of 30 seconds, followed by active stimulation with a steady current of two milliamps for 20 minutes, then a ramp-down of 30 seconds.
  Interventions: Device: tDCS; Behavioral: Cognitive Training
- Sham transcranial Direct Current Stimulation (tDCS) + Cognitive training (CT) (Sham Comparator): Twenty-three participants received five treatment sessions of concurrent sham tDCS and CT on five consecutive days. The current was only delivered in the 30-second ramp-up and 30-second ramp-down periods.
  Interventions: Device: tDCS; Behavioral: Cognitive Training

INTERVENTIONS:
Device: tDCS — tDCS was applied using the StarStim 8 (NeuroElectrics, Barcelona, Spain). tDCS with strength of two milliamps for 20 minutes was applied based on montage recommended (Hoy et al., 2014). The stimulation electrode was applied according to international EEG system 10-20. The anode was applied at the left dorsolateral prefrontal cortexDLPFC, which was located at F3; the cathode was applied at the right dorsolateral prefrontal cortexDLPFC, which was located at F4. In the tDCS group, the participants received 'ramp-up' of 30 seconds, followed by active stimulation with a steady current of two milliamps for 20 minutes, then 'ramp-down' of 30 seconds. In the sham group, the current was only delivered in the 30-second 'ramp-up' and 30-second 'ramp-down' period.
  Other Names: StarStim 8
Behavioral: Cognitive Training — All participants received the same program of cognitive training in the app 'the Peak' on a hand-held portable iPad (https://www.peak.net/science/). The traditional Chinese version with Cantonese instructions was selected. The progress, the errors, and the sum scores were stored in the personal profile for interactive feedback on adjusting the difficulty level. The participants performed the tasks in pseudorandomized order during each session. Each training session lasted for 20 minutes, concurrent with either active or sham tDCS stimulation.

SUMMARY:
Given the superior effects of CT augmented tDCS in healthy subjects, the aim of the current study was to examine whether the effect of CT on cognition can be enhanced with concurrent anodal tDCS in schizophrenia patients. A double-blinded randomised controlled trial design was utilised and cognitive performances were examined at baseline (T0), immediately after the intervention (T1) and one month post-intervention (T2). It was hypothesized that concurrent CT with tDCS would result in greater and more sustainable cognitive improvement than CT alone because of increased susceptibility to neuroplasticity changes of the underlying activated network (Bikson et al., 2013; Orlov, O'Daly, et al., 2017). The effects of concurrent CT with tDCS were also assessed using blinded assessments of psychotic, negative symptoms, affective symptoms, psychosocial functioning, subjective quality of life (QOL) and tolerability in the two groups.

DETAILED DESCRIPTION:
The current study is a parallel-group, double-blinded, randomised controlled trial that aimed to fill the knowledge gap in investigating the effect of five sessions of concurrent cognitive training with 'online' tDCS on specific cognitive domains in stable schizophrenia patients at two time-points, (i) immediately after the intervention (ii) at one month after intervention.

It was hypothesized that concurrent cognitive training with 'online' tDCS would result in greater incremental effective improvements in cognitive domains as compared to the cognitive training alone, and the effect would be sustainable at one-month follow-up. The effect of the concurrent cognitive training with 'online' tDCS were also assessed using blinded assessments of psychotic, negative symptoms, affective symptoms, psychosocial functioning, subjective quality of life (QOL) and tolerability in the two groups.

Participant were randomly allocated to one of the two groups using a predetermined randomisation sequence and block randomisation generator (block of 6). Group 1 received active tDCS stimulation and CT and will be referred to as the active tDCS + CT group. Group 2 received sham tDCS and CT and will be referred to as the sham tDCS + CT group. Both groups consisted of 23 participants and received five treatment sessions on five consecutive days.

Stimulation protocol with the corresponding randomisation code was set up by an independent psychiatrist.The double-blind administration panel of the SatrStim8 system of tDCS ensured effective blinding; both the principal investigator and the participants were blinded to the group allocation until the statistical analysis stage. All outcome measures were assessed at three time-points (T0, baseline; T1, end-treatment course; and T2, at one-month post-intervention).

Declaration:

The research protocol fully complies with the Declaration of Helsinki and the guidelines of ICH-GCP.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18-65 years old; and
2. Being right handed; and
3. Able to communicate in Cantonese; and
4. With the diagnosis of schizophrenia meeting the diagnostic criteria of the World Health Organization's 10th version of the International Statistical Classification of Disease and Related Health Problems (ICD-10). All diagnoses were ascertained at multidisciplinary team and endorsed by at least a consultant psychiatrist and a specialist in psychiatry in the clinical teams based in Tai Po Hospital.

Exclusion Criteria:

1. Significant neurologic history such as dementia, stroke, seizure, Parkinson's disease, multiple sclerosis; or
2. History of brain neurosurgery; or
3. Active abuse of alcohol or illicit substances; or
4. Concurrent use of cognitive-enhancing medications e.g. acetylcholinesterase inhibitors; or
5. Documented history of learning disability; or
6. Implanted with pacemakers, intracranial electrodes, defibrillators, metal implants in head or neck area; or
7. Pregnancy or breastfeeding; or
8. Changes in medication regime over the two weeks before or during the study period (Brunoni, Ferrucci, et al., 2011).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Cambridge Neuropsychological Test Automated Battery | Score change baseline versus post-intervention versus week 4
  After a first touch screen adaption period, the participants performed four CANTAB tasks always in the same order: Reaction Time (RTI - Simple and Five choice Tone), Paired Associates Learning (PAL - Recommended Standard), Spatial Working Memory (SWM - Recommended Standard 2.0) and Rapid Visual Information Processing (RVP).The key variables from each CANTAB task were selected as the a priori primary measures.
Trail Making Test, Part A | Score change baseline versus post-intervention versus week 4
  Part of the MCCB measure and has a brief administration time, high tolerability, good test-retest reliability and potential changeability in response to pharmacological agents (Nuechterlein et al., 2008).
Backward Digit Span | Score change baseline versus post-intervention versus week 4
  The test was administered according to the instructions provided in the WAIS-IV-HK administration manual. A list of digits at a rate of one per second was read aloud, and the list was repeated in the reverse order to presentation order. All digits must be in the correct order for the list to be marked correct. The list started at a length of two digits, and two lists of each length were read aloud. The maximum span length correctly recalled was selected as the primary measure of the maximum capacity of the participant's working memory.

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale | Score change baseline versus post-intervention versus week 4
  It is a 30-item clinician rated questionnaire to assess the symptoms in schizophrenia patient. It has three sub-categories of positive symptoms, negative symptoms and general psychopathology. It is shown to have good construct validity , internal reliability and inter-rater reliability (Lindstrom et al., 1994). It is also shown to be sensitive to change (Santor et al., 2007). Each item is rated on a 7-point scale. Minimum value is 30 and maximum value is 210. Higher score indicates more severe symptoms.
Calgary Depression Scale for Schizophrenia (CDSS) | Score change baseline versus post-intervention versus week 4
  It is a nine-item clinician rated questionnaire. It is administered following a semi-structured interview. It has been used by other tDCS studies in schizophrenia, and it has been shown to be reliable, valid and sensitive to depressive symptoms separate from positive, negative and extrapyramidal symptoms in schizophrenia. A score above six has 82% specificity and 85% sensitivity for predicting the presence of a major depressive episode
Clinical Global Impression Scale | Score change baseline versus post-intervention versus week 4
  It is a three-item clinician rated questionnaire to assess illness severity, global improvement or change, and treatment response. Higher scores indicate more severe pathology. The first two items can be rated from 1-7 and the third item consist of a 4×4 rating scale (1-16) that assesses the therapeutic effect of treatment and associated side effects.
Social and Occupational Functioning Assessment scale (SOFAS) | Score change baseline versus post-intervention versus week 4
  It is a 100-point single-item rating scale to assess patients' personal and social functioning. A score of 0 indicates "Inadequate information". A score of 10 indicates Persistent inability to maintain minimal personal hygiene. Unable to function without harming self or others or without considerable external support (e.g., nursing care and supervision), while a score of 100 indicates superior functioning in a wide range of activities.
World Health Organization Five Well-Being Index (WHO-5) | Score change baseline versus post-intervention versus week 4
  It is a five-item self-reported questionnaire of subjective quality of life.
Ratings on Motivation and Enjoyment on Cognitive Training. | Score change baseline versus post-intervention versus week 4
  Visual Analog Scale to rate their motivation and enjoyment to participate in the gamified computerised cognitive training programme (scores ranged from 0-100, with higher scores indicating enhanced enjoyment/ willingness to come).
An Adverse Effects Questionnaire | Score change baseline versus post-intervention versus week 4
  It is associated with tDCS administration, which has been generated from a systematic review in 2011 by Brunoni.
Beck Cognitive Insight Scale Taiwanese Version | Score change baseline versus post-intervention versus week 4
  It is 15-tem self-reported questionnaire with two subscales (nine items tapping self-reflectiveness and six on self-certainty). It is shown to have Cronbach's alpha values of >0.70 for both subscales and has moderate stability.

CONTACTS AND LOCATIONS:
Overall Officials: Ka Ying Heidi Lo, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Psychiatry, CUHK, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
As they are all clinical subjects, their data should be strictly confidential.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/96/NCT04870996/Prot_SAP_000.pdf